CLINICAL TRIAL: NCT04986319
Title: The Level of Serum Vitamin D And Parathyroid Hormone Among Different Bangladeshi Population Groups
Brief Title: Reference Interval of Vitamin D of Coastal Fishermen in Cox's Bazar District of Bangladesh
Status: Completed | Type: Observational
Sponsor: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (Other)
Collaborators: Bangladesh Medical Research Council (BMRC) (Other)
Responsible Party: Principal Investigator, Wasim Md Mohosin Ul Haque, Associate Professor, Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders
Other Study IDs: BADAS-ERC/EC/21/00310
Record Dates: First submitted 2021-05-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Bangladesh; Optimal Level; Coastal fishermen; Parathyroid Hormone; Reference interval
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adequately sun-exposed healthy population: Healthy coastal fishermen of Cox's Bazar district of Bangladesh
  Interventions: Diagnostic Test: Serum vitamin D assay
- Inadequately sun-exposed healthy population: Healthcare workers of the selected hospitals of Dhaka, Bangladesh
  Interventions: Diagnostic Test: Serum vitamin D assay

INTERVENTIONS:
Diagnostic Test: Serum vitamin D assay — Trained phlebotomists will collect 10 cc of a Blood sample. Specimen will be preserved at -40ºc for batch analysis.
  S Vitamin D, S iPTH, S Calcium, S Alkaline Phosphatase, S PO4, S Mg, S Albumin and S Creatinine will be done in BIRDEM laboratory. Vitamin D will be assayed by The ARCHITECT 25-OH Vitamin D assay system: Vitamin D will be assayed by The ARCHITECT 25-OH Vitamin D assay system: The ARCHITECT 25-OH Vitamin D assay is a chemiluminescent micro-particle immunoassay (CMIA). This technology is used for the quantitative analysis of 25(OH) D and aid in the assessment of vitamin D sufficiency.
  Other Names: Serum iPTH assay

SUMMARY:
Lack of adequate sun exposure due to urbanization is prone to hypovitaminosis D. Vitamin D (25-hydroxyvitamin D) deficiency is now a major health concern in the western world. Recent data suggest that Vitamin D level in the Bangladeshi population is also very low. However, the cutoff value used to determine vitamin D deficiency is not yet validated for our ethnic group; we also don't know the optimal vitamin D level for our population. Before coming to any firm conclusion regarding nationwide vitamin D deficiency, we must know the Optimal range of serum Vitamin D for our people of Bangladesh. As sunlight is the primary source of vitamin D and adequate sun exposure alone is sufficient to produce enough vitamin D to maintain the physiological demand without producing toxicity. According to Holick's rule, exposure to sunlight at the face and both arms for 25 min, 3 times a week should maintain adequate vitamin D status. In Indonesia, it was found that after exposure to sunlight at this specific time and duration for 6 weeks, the mean 25(OH)D levels of participants increased from 59 nmol/L at the baseline to 84 nmol/L.In India, exposure to sunlight for 30 minutes, between 11 am and 2 pm, three times a week, is sufficient to maintain adequate serum vitamin D concentration. Therefore it could be assumed that healthy subjects without any risk factors for vitamin D deficiency and having adequate sun exposure should maintain an Optimal serum vitamin D concentration. Here Optimal means a range where there will be no features of insufficiency or toxicity. In this cross-sectional study, we want to find out the serum vitamin D level of such a population, representing the Optimal level of vitamin D for Bangladeshi people.

DETAILED DESCRIPTION:
Vitamin D is the sunshine vitamin produced on this earth for more than 500 million years. This is produced in humans by sunlight. Sunlight is the main source of vitamin D, and adequate sun exposure alone is sufficient to produce enough vitamin D to maintain the physiological demand without producing toxicity. According to Holick's rule, exposure to sunlight on the face and both arms for 25 min, 3 times a week, should maintain adequate vitamin D status. In Indonesia, it was found that after exposure to sunlight at this specific time and duration for 6 weeks, the mean 25(OH)D levels of participants increased from 59 nmol/L at the baseline to 84 nmol/L.In India, exposure to sunlight for 30 minutes, between 11 am and 2 pm, three times a week is sufficient to maintain adequate serum vitamin D concentration. Lack of adequate sun exposure as a consequence of urbanization prone human races to a threat of hypovitaminosis D. Vitamin D (25-hydroxyvitamin D) insufficiency and its impending consequence on health is now the subject of important concern and controversy. The optimal value of vitamin D substantially differs among populations depending upon environmental, cultural and racial factors. However, the definition of vitamin D insufficiency is still not out of controversy, mostly cutoffs of <50 nmol/L of serum 25-hydroxyvitamin D (25(OH)D) level is considered as "vitamin D deficiency" state, 50 to 74.9 nmol/L denotes "insufficiency" and ≥75 nmol/L considered as "sufficiency".

With the falling of serum25 (OH)D beyond a certain point, absorption of calcium from the gut decreases, which leads to a surge of parathyroid hormone (PTH) secretion, which in turn stimulates the conversion of 25(OH)D to 1,25(OH)2D to keep calcium at a normal limit. Thus, a higher value of PTH could be considered as a surrogate marker of vitamin D insufficiency. Serum 25(OH) D below the level of 75-100 nmol/L has an inverse correlation with PTH concentration; beyond this point, serum intact PTH concentration remains in a plateau state.

Based on these definitions, the whole world faces a pandemic of vitamin D deficiency/insufficiency. According to recent studies, the prevalence of vitamin D deficiency has been found between 30% and 100% in different communities. This picture is similar in the USA, Europe, South East Asia and the Middle East. In India, the prevalence of Vitamin D deficiency is around 70%-100% in the general population. Baidya et al. (2012) studied 40 healthy Indian physicians in Calcutta. Around 97.5% of subjects had low vitamin D. Mean age and meant 25(OH)D levels of that cohort were 52.22 ± 10 years and 13.02 ± 4.77 ng/ml (32.50±11.91 nmol/L). Vitamin D deficiency was found in 92.5% of participants. Though available data in Bangladesh are confined to female subjects only, the scenario is not different. More than ninety-nine percent of Bangladesh female garment workers were vitamin D insufficient in a study.

This picture is alarming because, in addition to its deleterious effect on the musculoskeletal system, vitamin D deficiency is also linked with many other medical issues like cardiovascular disease, malignancy, neuromodulation, diabetes, and metabolic syndrome several autoimmune diseases (such as multiple sclerosis, Crohn's disease and ulcerative colitis) and certain infectious diseases, such as tuberculosis. Vitamin D supplementation is also a key component in the hierarchy of management of Chronic Kidney Disease-Mineral and Bone Disorder.

However, the caveat of all of those studies done in Bangladesh and neighbouring countries like India and Pakistan is that the cutoff value used to determine vitamin D deficiency or insufficiency has not yet been validated for the corresponding population. Before reaching a firm conclusion about epidemics of vitamin D deficiency and planning for supplementation programs, the cutoff value of vitamin D deficiency/insufficiency of the Bangladeshi population must be validated. The optimal level of vitamin D for the Bangladeshi population should also find out.

Rationale: Maintenance of adequate vitamin D levels undoubtedly is an important human health issue. It helps prevent many chronic diseases, which in fact are in addition to its principal role in maintaining appropriate blood calcium levels. To get the optimum beneficial effects of vitamin D, including prevention of many potential adverse health effects caused by deficient vitamin D, circulating 25(OH)D levels should be within the normal range. Vitamin D varies depending on various factors like exposure to the sun, age, race, body mass index, lack of exercise etc. The cutoff value for deficiency and insufficiency also varies between studies. Several studies using prescribed cutoff values of vitamin D deficiency reveal an epidemic of vitamin D deficiency in our country, despite abounded sunlight due to the proximity of the equator. However, no study was done previously in Bangladesh to determine the Optimal value of vitamin D representative of this population. The deficiency and insufficiency levels are ignorant and when to intervene is also not known. That is why it is important to conduct this exploratory study. It will help to assume the optimal reference range of serum vitamin D for the Bangladeshi population. That will give a clearer picture of the actual burden of vitamin D deficiency in Bangladesh and guide them to treat them and take necessary preventive measures at the national level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy fishermen
* Healthy health care workers
* Who will be willing to participate in the study

Exclusion Criteria:

* Those who will refuse to participate in the interview
* Physically and psychologically handicapped
* Subjects with known chronic illnesses like liver, kidney or gastrointestinal disease, metabolic bone disease, malignancy, pregnancy and lactation, history of immobility for more than 1 week, on vitamin D or calcium supplementation, on anti-epileptic drugs
* Primary hyperparathyroidism
* Subject having lactose intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adequately sun-exposed healthy population: Healthy fishermen with at least 30 minutes of sun exposure between 11 am and 2 pm, three times a week for the preceding 6 months.
  All male aged 18 to 65 years
  Inadequately sun-exposed healthy population: Urban, office-based workers or homemakers, both male and female, who will come for a routine health check-up in the BIRDEM outpatient department, and health care workers of selected hospitals of Dhaka. Both male and female aged 18 to 65 years.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D levels | Day 1
  Serum vitamin D levels of healthy fishermen, healthy volunteers and healthy healthcare workers will be measured in the chemiluminescent microparticle immunoassay method.

SECONDARY OUTCOMES:
Serum parathyroid hormone levels | Day 1
  Serum parathyroid hormone levels of healthy fishermen, healthy volunteers and healthy healthcare workers will be measured in the chemiluminescent microparticle immunoassay method.

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Md Mohosin Ul Haque, FCPS, Principal Investigator — Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders
Locations (2):
- Bangladesh (2):
  - Cox's Bazar, Cox’s Bāzār
  - BIRDEM General Hospital, Dhaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wacker M, Holick MF. Sunlight and Vitamin D: A global perspective for health. Dermatoendocrinol. 2013 Jan 1;5(1):51-108. doi: 10.4161/derm.24494. PMID 24494042
- [Background] Nimitphong H, Holick MF. Vitamin D status and sun exposure in southeast Asia. Dermatoendocrinol. 2013 Jan 1;5(1):34-7. doi: 10.4161/derm.24054. PMID 24494040
- [Background] Harinarayan CV, Holick MF, Prasad UV, Vani PS, Himabindu G. Vitamin D status and sun exposure in India. Dermatoendocrinol. 2013 Jan 1;5(1):130-41. doi: 10.4161/derm.23873. PMID 24494046
- [Background] Holick MF. Sunlight and vitamin D for bone health and prevention of autoimmune diseases, cancers, and cardiovascular disease. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1678S-88S. doi: 10.1093/ajcn/80.6.1678S. PMID 15585788
- [Background] Walentowicz-Sadlecka M, Sadlecki P, Walentowicz P, Grabiec M. [The role of vitamin D in the carcinogenesis of breast and ovarian cancer]. Ginekol Pol. 2013 Apr;84(4):305-8. doi: 10.17772/gp/1581. Polish. PMID 23700865
- [Background] Wacker M, Holick MF. Vitamin D - effects on skeletal and extraskeletal health and the need for supplementation. Nutrients. 2013 Jan 10;5(1):111-48. doi: 10.3390/nu5010111. PMID 23306192
- [Background] Wimalawansa SJ. Vitamin D in the new millennium. Curr Osteoporos Rep. 2012 Mar;10(1):4-15. doi: 10.1007/s11914-011-0094-8. PMID 22249582
- [Background] Holick MF. Vitamin D: extraskeletal health. Rheum Dis Clin North Am. 2012 Feb;38(1):141-60. doi: 10.1016/j.rdc.2012.03.013. Epub 2012 Apr 12. PMID 22525849
- [Background] Bischoff-Ferrari H. Vitamin D - from essentiality to functionality. Int J Vitam Nutr Res. 2012 Oct;82(5):321-6. doi: 10.1024/0300-9831/a000126. PMID 23798050
- [Background] Moreno LA, Valtuena J, Perez-Lopez F, Gonzalez-Gross M. Health effects related to low vitamin D concentrations: beyond bone metabolism. Ann Nutr Metab. 2011;59(1):22-7. doi: 10.1159/000332070. Epub 2011 Nov 25. PMID 22123633
- [Background] Need AG, Horowitz M, Morris HA, Nordin BC. Vitamin D status: effects on parathyroid hormone and 1, 25-dihydroxyvitamin D in postmenopausal women. Am J Clin Nutr. 2000 Jun;71(6):1577-81. doi: 10.1093/ajcn/71.6.1577. PMID 10837301
- [Background] von Muhlen DG, Greendale GA, Garland CF, Wan L, Barrett-Connor E. Vitamin D, parathyroid hormone levels and bone mineral density in community-dwelling older women: the Rancho Bernardo Study. Osteoporos Int. 2005 Dec;16(12):1721-6. doi: 10.1007/s00198-005-1910-8. Epub 2005 Jun 1. PMID 15928802
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Thomas MK, Lloyd-Jones DM, Thadhani RI, Shaw AC, Deraska DJ, Kitch BT, Vamvakas EC, Dick IM, Prince RL, Finkelstein JS. Hypovitaminosis D in medical inpatients. N Engl J Med. 1998 Mar 19;338(12):777-83. doi: 10.1056/NEJM199803193381201. PMID 9504937
- [Background] Chapuy MC, Preziosi P, Maamer M, Arnaud S, Galan P, Hercberg S, Meunier PJ. Prevalence of vitamin D insufficiency in an adult normal population. Osteoporos Int. 1997;7(5):439-43. doi: 10.1007/s001980050030. PMID 9425501
- [Background] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Background] Vierucci F, Del Pistoia M, Fanos M, Erba P, Saggese G. Prevalence of hypovitaminosis D and predictors of vitamin D status in Italian healthy adolescents. Ital J Pediatr. 2014 Jun 5;40:54. doi: 10.1186/1824-7288-40-54. PMID 24902694
- [Background] G R, Gupta A. Vitamin D deficiency in India: prevalence, causalities and interventions. Nutrients. 2014 Feb 21;6(2):729-75. doi: 10.3390/nu6020729. PMID 24566435
- [Background] Beloyartseva M, Mithal A, Kaur P, Kalra S, Baruah MP, Mukhopadhyay S, Bantwal G, Bandgar TR. Widespread vitamin D deficiency among Indian health care professionals. Arch Osteoporos. 2012;7:187-92. doi: 10.1007/s11657-012-0096-x. Epub 2012 Sep 28. PMID 23225296
- [Background] Zargar AH, Ahmad S, Masoodi SR, Wani AI, Bashir MI, Laway BA, Shah ZA. Vitamin D status in apparently healthy adults in Kashmir Valley of Indian subcontinent. Postgrad Med J. 2007 Nov;83(985):713-6. doi: 10.1136/pgmj.2007.059113. PMID 17989271
- [Background] Isaia G, Giorgino R, Rini GB, Bevilacqua M, Maugeri D, Adami S. Prevalence of hypovitaminosis D in elderly women in Italy: clinical consequences and risk factors. Osteoporos Int. 2003 Jul;14(7):577-82. doi: 10.1007/s00198-003-1390-7. Epub 2003 Jul 11. PMID 12856111
- [Background] Sedrani SH. Low 25-hydroxyvitamin D and normal serum calcium concentrations in Saudi Arabia: Riyadh region. Ann Nutr Metab. 1984;28(3):181-5. doi: 10.1159/000176801. PMID 6610383
- [Background] Goswami R, Gupta N, Goswami D, Marwaha RK, Tandon N, Kochupillai N. Prevalence and significance of low 25-hydroxyvitamin D concentrations in healthy subjects in Delhi. Am J Clin Nutr. 2000 Aug;72(2):472-5. doi: 10.1093/ajcn/72.2.472. PMID 10919943
- [Background] Hwang JS, Tsai KS, Cheng YM, Chen WJ, Tu ST, Lu KH, Hou SM, Yang SH, Cheng H, Lai HJ, Lei S, Chen JF. Vitamin D status in non-supplemented postmenopausal Taiwanese women with osteoporosis and fragility fracture. BMC Musculoskelet Disord. 2014 Jul 28;15:257. doi: 10.1186/1471-2474-15-257. PMID 25069806
- [Background] Baidya A, Chowdhury S, Mukhopadhyay S, Ghosh S. Profile of vitamin D in a cohort of physicians and diabetologists in Kolkata. Indian J Endocrinol Metab. 2012 Dec;16(Suppl 2):S416-7. doi: 10.4103/2230-8210.104113. PMID 23565448
- [Background] Micka A. Vitamin D Status among Bangladeshi Women of Reproductive Age [Masters Theses ]. ScholarWorks@UMass Amherst: University of Massachusetts Amherst; 2009
- [Background] Islam MZ, Lamberg-Allardt C, Karkkainen M, Outila T, Salamatullah Q, Shamim AA. Vitamin D deficiency: a concern in premenopausal Bangladeshi women of two socio-economic groups in rural and urban region. Eur J Clin Nutr. 2002 Jan;56(1):51-6. doi: 10.1038/sj.ejcn.1601284. PMID 11840180
- [Background] Islam MZ, Akhtaruzzaman M, Lamberg-Allardt C. Hypovitaminosis D is common in both veiled and nonveiled Bangladeshi women. Asia Pac J Clin Nutr. 2006;15(1):81-7. PMID 16500882
- [Background] Islam MZ, Shamim AA, Kemi V, Nevanlinna A, Akhtaruzzaman M, Laaksonen M, Jehan AH, Jahan K, Khan HU, Lamberg-Allardt C. Vitamin D deficiency and low bone status in adult female garment factory workers in Bangladesh. Br J Nutr. 2008 Jun;99(6):1322-9. doi: 10.1017/S0007114508894445. PMID 18430266
- [Background] Roth DE, Shah MR, Black RE, Baqui AH. Vitamin D status of infants in northeastern rural Bangladesh: preliminary observations and a review of potential determinants. J Health Popul Nutr. 2010 Oct;28(5):458-69. doi: 10.3329/jhpn.v28i5.6154. PMID 20941897
- [Background] Ketteler M, Block GA, Evenepoel P, Fukagawa M, Herzog CA, McCann L, Moe SM, Shroff R, Tonelli MA, Toussaint ND, Vervloet MG, Leonard MB. Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder: Synopsis of the Kidney Disease: Improving Global Outcomes 2017 Clinical Practice Guideline Update. Ann Intern Med. 2018 Mar 20;168(6):422-430. doi: 10.7326/M17-2640. Epub 2018 Feb 20. PMID 29459980